CLINICAL TRIAL: NCT01745484
Title: Role of SPECT in Radiotherapy Treatment Planning and Toxicity Evaluation for the Patients With Stage I-III NSCLC
Brief Title: Role of SPECT in Radiotherapy of Lung Cancer and Toxicity Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Katherina Farr, Principle Investigator, University of Aarhus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KFE-1203
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Non-small-cell Lung Cancer; Radiation Pneumonitis
Keywords: SPECT; Toxicity; Non-small-cell lung cancer; Definitive Radiotherapy; Radiation pneumonitis; Randomized study
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Radiation Pneumonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): SPECT scan will be performed at baseline. Patients will receive radiotherapy according to standard CT-based plan with conventional dose-volume histogram
  Interventions: Other: SPECT-based treatment plan

INTERVENTIONS:
Other: SPECT-based treatment plan — SPECT will be performed on all patients at baseline. Two treatment plans will be made- functional SPECT-based plan and conventional CT-based plan. Randomization will take place if both plans are satisfying established criteria for tumour coverage and normal tissue sparing. Randomization between Arm 1 and Arm 2 will be done, where the patients will be treated either by SPECT-plan or by CT-plan respectively.
  The SPECT data are viewed as a multicoloured image in the spectrum colour setting to allow accurate volume contouring around a predefined colour. The threshold level is adjusted individually for each patient in order to match the size of the SPECT image within the lung volumes defined on CT. A new contour of functional lung is created from the SPECT images using a threshold of 30% of the maximum uptake for each patient. A treatment plan is generated. The principal objective for each plan is to minimize the volume of lungirradiated
  Other Names: Single Photon Emission Computed Tomography

SUMMARY:
Overall objective of the study is to compare the use of SPECT in radiotherapy treatment planning with standard CT-based radiotherapy for stage I-III non-small-cell lung cancer patients

DETAILED DESCRIPTION:
Primary objective:

-To compare the rate of grade 2 or higher pneumonitis amongst patients with stage III NSCLC treated with radiotherapy using SPECT in radiotherapy treatment planning versus standard CT-based radiotherapy planning;

Secondary Objectives:

* To evaluate SPECT as a tool to predict lung toxicity;
* To establish estimates for the incidence and severity of pulmonary tissue effects observed in stage III NSCLC patients treated with radiotherapy;
* To generate hypotheses for subsequent use of SPECT-CT-based treatment planning as a method for minimization of toxicity risks
* To generate hypotheses for modeling studies of SPECT-CT-based treatment planning for dose-escalation;
* To compare the loco-regional control, time to progression and overall survival of patients treated with SPECT-based plan versus standard CT-based plan
* To compare the quality of life in patients randomized to the two study arms.

This trial is a single centre observational study. All patients will irrespective of their registration in the trial receive radiotherapy according to the standard treatment regimen at the Department of Oncology, Aarhus University Hospital. Participation implies baseline and follow-up procedures. In the treatment planning phase patients will be randomized to one of the following arms: Arm 1 SPECT/CT-based treatment plan with functional dose-volume parameters and Arrm 2 Standard CT-based plan with conventional dose-volume parameters.

The trial will consist of two parts. To initiate the trial a pilot study (part 1) will be performed to determine the feasibility in our setting at Aarhus University Hospital as it is described in the literature. Consecutive patients will be enrolled in the pilot study during 1-year period. The interim analysis after one year of enrollment will be performed to determine what patients are most likely to benefit from functional radiotherapy planning based on SPECT. The main objective of this part is to determine whether V/Q-SPECT data are valid and usable in the radiotherapy planning. The timing for acute and late follow-up SPECT will be determined. Randomized trial (part 2) will be performed thereafter.

Statistical analysis. The randomization by permitted blocks method will be used to allocate patients to treatment arm. Stratification factors will be age, gender, disease stage, histology, concurrent chemotherapy and irradiated volumes.

The chi-squire test (α=0.10) with the continuity correction will be used for analysis of the primary analysis. For all other comparisons, two-sided analyses will be performed and a p-value of 0.05 or less will be considered statistically significant. 95% confidence intervals will be constructed for outcomes of interest. Descriptive statistics will be used to summarize patient characteristics and outcomes by intervention arm. Differences in outcomes between intervention arms will be compared by using paired t-tests, Wilcoxon rank sum tests or McNemar tests as appropriate. Adjusting for stratification factors will be performed using logistic regression or linear regression. Time-to-event analyses will be estimated using the Kaplan-Meier method, and compared using Cox proportional hazards regression.

Estimation of the relationship between dose-volume parameters and toxicity will be evaluated using logistic regression analyses. Within patients who were planned using SPECT, the association between dose-volume parameters calculated using SPECT and those calculated under a CT-plan will be evaluated using correlation coefficients.

All patients who are randomized will be included in the analysis of safety and efficacy outcomes. Secondary analyses may be performed on those patients only on those who received radiotherapy as per the treatment plan based on SPECT or CT as per the intervention arm. Any patient who is randomized but does not receive radiotherapy based on the intervention allocated treatment plan will be described in detail along with the reason for not receiving the prescribed plan.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III non-small cell lung cancer, histologically verified
* Referred for definitive radiotherapy to the Department of Oncology, Aarhus University Hospital
* Meet the criteria for curatively intended radiotherapy described in details in the national guidelines
* Concurrent chemotherapy is accepted
* Adults over 18, that have given oral and written informed consent before patient registration
* The patients can only be randomized in this trial once

Exclusion Criteria:

* other uncontrolled malignancies
* human albumin allergy
* any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Grade 2 radiation pneumonitis | measured 0-12 months after completed radiotherapy
  The primary endpoint is grade 2 pneumonitis, defined according to the NCI Common Toxicity Criteria for Adverse Events (CTC) version 4.0.
  Estimation of the occurrence of pulmonary tissue effects:
  Number of patients developing pulmonary toxicity over grade 2 in both treatment arms according to the Common Terminology Criteria for Adverse Events CTC v. 4.0 and measured serially from 0 to 12 months after radiotherapy, as well as according to the SOMA-LENT scale measured serially from 0 to 12 months after radiotherapy

SECONDARY OUTCOMES:
Overall quality of life score | 0-12 months after radiotherapy
  Change in quality of life according to the standard quality of life questionnaires
Mean lung dose (MLD) and V5-50(volume of the lung receiving 5-50 Gy or more) | 12 months after radiotherapy
  Estimation of conventional (from CT alone) and functional (from SPECT)dose-volume parameters (MLD and V5-50) and their correlation with pulmonary toxicity will be done.
Progression-free survival | at 12 months after radiotherapy
  Proportion of patients alive with no evidence of disease as per the RECIST criteria in the SPECT arm compared to CT arm

CONTACTS AND LOCATIONS:
Overall Officials: Katherina Farr, MD, Principal Investigator — Department of Oncology, Aarhus University Hospital
Locations (1):
- Department of Oncology, Aarhus University Hospital, Aarhus, Denmark